CLINICAL TRIAL: NCT00072189
Title: A Phase II Study of UCN-01 in Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination for discouraging results
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02829; NCI-2012-02829 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-33 (Other: City of Hope); 5536 (Other: CTEP); N01CM17101 (NIH)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — 7-hydroxystaurosporine

ARMS (1):
- Treatment (7-hydroxystaurosporine) (Experimental): Patients receive UCN-01 IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 7-hydroxystaurosporine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: 7-hydroxystaurosporine — Given IV
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies

SUMMARY:
UCN-01 may stop the growth of tumor cells by blocking the enzymes necessary for their growth. This phase II trial is studying how well UCN-01 works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the anti-tumor activity of UCN-01 (7-hydroxystaurosporine) in metastatic melanoma, as determined by the response rate.

II. To assess the clinical and laboratory toxicities of UCN-01. III. To study the effects of UCN-01 administration on potential markers of specific G1-phase cell cycle regulators.

OUTLINE: This is a multicenter study.

Patients receive UCN-01 IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 17-33 patients will be accrued for this study within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients have histologically or cytologically confirmed melanoma that is incurable by other means such as surgery, radiotherapy, or limb perfusion
* Patients must have measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with conventional techniques or with spiral CT scan, and which has clearly progressed during the observation interval prior to participation in this study
* Patients must have received =< 1 prior chemotherapy and/or =< biological therapies; isolated limb perfusion with a biological and/or chemotherapeutic agent is allowed if the measurable disease and the lesion that will be biopsied for this protocol are outside the area of prior perfusion; at least 4 weeks must have elapsed since prior therapy (6 weeks for nitrosoureas or mitomycin C) and the patient must have recovered from all toxicities attributable to prior therapy
* Life expectancy greater than 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status #2 (Karnofsky >= 60%)
* Leukocytes >= 3000/uL
* Absolute neutrophil count >= 1500/uL
* Platelets >= 100000/uL
* Total bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 X institutional upper limit of normal
* Creatinine < 1.6 mg/dL
* Creatinine clearance >= 50 mL/min for patients with creatinine levels above 1.6 mg/dL
* The effects of UCN-01 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign a written informed consent document
* Patient must have a central venous catheter
* Patients are requested to submit archival tissue for pre-study and undergo a tumor biopsy 24 hours post UCN-01 administration if feasible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or who have not recovered from adverse events to agents administered more than 4 weeks earlier
* Patients must not be receiving any other investigational agents
* Patients with known brain metastases are eligible only if disease is controlled and patient is asymptomatic (i.e. at least 4 weeks from completion of whole brain irradiation, stereotactic radiosurgery, or gamma knife irradiation) and not receiving corticosteroids
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to UCN-01
* Patients with only non-measurable disease, defined as all other lesions, including small lesions (longest diameter >= 10 mm with conventional techniques or with spiral CT scan) and truly non-measurable lesions, which include the following:

  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural or pericardial effusion
  * Abdominal masses that are not confirmed and followed by imaging techniques
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, systematic congestive heart failure, symptomatic pulmonary diseases, unstable angina pectoris, cardiac arrhythmia, prior mediastinal radiation or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because UCN-01 is a serine-threonine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse effects in nursing infants secondary to treatment of the mother with UCN-01, breastfeeding should be discontinued if the mother is treated with UCN-01
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with UCN-01; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Due to the incidence of hyperglycemia with UCN-01, patients with a history of diabetes will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Christensen, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- [Derived] Li T, Christensen SD, Frankel PH, Margolin KA, Agarwala SS, Luu T, Mack PC, Lara PN Jr, Gandara DR. A phase II study of cell cycle inhibitor UCN-01 in patients with metastatic melanoma: a California Cancer Consortium trial. Invest New Drugs. 2012 Apr;30(2):741-8. doi: 10.1007/s10637-010-9562-8. Epub 2010 Oct 22. PMID 20967484

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Patients receive UCN-01 IV at 90 mg/m2 over 3 hours on cycle 1, reduced to 45 mg/m2 over 3 hours for subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  7-hydroxystaurosporine: Given IV
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Period: Overall Study
Arm/Group | Arm 1
Started | 17
Completed | 16
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 53 [34 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 7 years
Measure: Number; unit: percentage of responding participants
Arm/Group | Arm 1
Number analyzed (Participants) | 16
percentage of responding participants | 0

2. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 17
months | 7.3 [3.4 to 18.4]

3. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of study registration to the first documentation of progressive tumor, assessed up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1
Number analyzed (Participants) | 17
months | 1.3 [1.2 to 3.0]

ADVERSE EVENTS:
Time Frame: Collected over a period of 24 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
General symptom (General disorders) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (16)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 1 (5)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (12)
Vomiting (Gastrointestinal disorders) | 6 (7)
Fatigue (General disorders) | 11 (25)
Fever (General disorders) | 1 (1)
General symptom (General disorders) | 7 (7)
Oedema NOS (General disorders) | 2 (2)
Pain (General disorders) | 2 (4)
Infection NOS (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 4 (7)
Creatinine increased (Investigations) | 4 (5)
Hyperbilirubinemia (Investigations) | 2 (2)
Hypercholesterolemia (Investigations) | 5 (16)
Leukopenia (Investigations) | 3 (11)
Lymphopenia (Investigations) | 3 (13)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (31)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Study was terminated early after the first stage of a two-stage design, allowing for early termination for discouraging results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less